CLINICAL TRIAL: NCT03281174
Title: Phase IV, Open-labelled, Five-year Immune Persistence Study of Inactivated Enterovirus Type 71 (EV71) Vaccine
Brief Title: Five-year Immune Persistence Study of Inactivated Enterovirus Type 71 (EV71) Vaccine
Status: Completed | Type: Observational
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-EV71-4007
Record Dates: First submitted 2017-09-08; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Inactivated Enterovirus Type 71 (EV71) Vaccine; 5-year Immune Persistence
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The venous blood was collected for EV71 neutralizing antibody detection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EV71 vaccine group: The group which received two doses EV71 vaccine (400U/0.5ml) on day 0,28 in phase III clinical trial.
- Placebo group: The group which received two doses placebo (0U/0.5ml) on day 0,28 in phase III clinical trial.

SUMMARY:
The purpose of this study is to evaluate the 5-year Immune Persistence of Inactivated Enterovirus Type 71 (EV71) Vaccine manufactured by Sinovac (Beijing) Biotech Co., Ltd.

DETAILED DESCRIPTION:
The phase III, efficacy trial of inactivated vaccine (vero cell) against EV71 has completed on March 2013 in China,and a follow up study for phase III clinical trial has completed on March 2014.

On the basis of phase III, this study is the Phase IV, open-labelled research, in order to evaluate the 5-year immune persistence of EV71 vaccine.

ELIGIBILITY:
Inclusion Criteria:

In the prior phase III clinical trial, 10077 subjects in three counties (Ganyu, Sheyang and Taixing ) were enrolled ( Experimental group: 5044; Control group: 5043 ), with 1293 of them in immunogenicity subgroup (Experimental group: 648; Control group: 645). In Sheyang county, 3351 subjects were enrolled (Experimental group: 1676 ; Control group :1675) , with 435 of them in immunogenicity subgroup (Experimental group: 418 ; Control group :418).

The subjects in Sheyang immunogenicity subgroup with the following conditions were included in this study:

* Guardian(s) of the volunteer should be capable of understanding the written consent form, and such form should be signed before the infant being included into this study
* Received at least one injection of EV71 vaccine or the placebo in the phase III clinical trial
* Finished the blood sampling 64 months after the vaccination

Exclusion Criteria:

* Received extra EV71 vaccination after the phase III clinical trial
* Refused to join the study

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The studied subjects are infants aged 6-35 months old infants when enrolled into the phase III clinical trial, and they are children aged 6-8 years old five years after the EV71 vaccine /placebo injection.
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2017-05-21 (Actual); Study Completion 2017-05-21 (Actual)

PRIMARY OUTCOMES:
The seropositive rate of EV71 neutralizing antibody-1 | 5 years (64 months)
  Calculated based on the cutoff value of 1:8

SECONDARY OUTCOMES:
The seropositive rate of EV71 neutralizing antibody-2 | 5 years (64 months)
  Calculated based on the cutoff value of 1:16
The seropositive rate of EV71 neutralizing antibody-3 | 5 years (64 months)
  Calculated based on the cutoff value of 1:32
The GMT of EV71 neutralizing antibody | 5 years (64 months)
  The GMT of EV71 neutralizing antibody 64 months after the first dose injection

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Principal Investigator — Jiangsu Provicial Center for Disease Control and Prevention
Locations (1):
- Sheyang Center for Disease Control and Prevention, Yancheng, Jiangsu, China

REFERENCES:
- [Derived] Hu Y, Zeng G, Chu K, Zhang J, Han W, Zhang Y, Li J, Zhu F. Five-year immunity persistence following immunization with inactivated enterovirus 71 type (EV71) vaccine in healthy children: A further observation. Hum Vaccin Immunother. 2018 Jun 3;14(6):1517-1523. doi: 10.1080/21645515.2018.1442997. Epub 2018 Apr 11. PMID 29482422